CLINICAL TRIAL: NCT06704828
Title: An Open-label, Multi-center Phase II Study to Evaluate the Safety, Tolerablity, Pharmacokinetics, and Efficacy of SHR-4602 as Montherapy or in Combination With Other Anti-tumor Therapies in Sujbects With Advanced Solid Tumors
Brief Title: A Phase II Study of SHR-4602 as Montherapy or in Combination With Other Anti-tumor Therapies in Advanced Solid Tumors
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Hengrui Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHR-4602-202
Record Dates: First submitted 2024-11-22; First posted 2024-11-26 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Advanced Solid Tumors

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SHR-4602 (Experimental)
  Interventions: Drug: SHR-4602

INTERVENTIONS:
Drug: SHR-4602 — SHR-4602

SUMMARY:
The study is being conducted to evaluate the safety, tolerability, pharmacokinetics and efficacy of SHR-4602 as montherapy or in combination with other anti-tumor therapies in advanced solid tumors. To explore the reasonable dosage of SHR-4602 for advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. 18-80 years old;
2. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1;
3. Stage I: subjects with pathologically confirmed locally advanced unresectable or metastatic solid tumors, who have failed at least 1 line of standard treatment;
4. Provide archived or fresh tumor tissue；HER2 expression is required for subjects in Stage I;
5. At least one measurable lesion according to RECIST v1.1；
6. Expected survival ≥12 weeks
7. Good level of organ function；
8. Female subjects of childbearing potential must have a negative serum pregnancy test within 7 days prior to the first dose, be non-lactating. Male subjects whose partners are women of childbearing age and female subjects who are fertile must agree to avoid sperm or egg donation during the treatment period until 8 months after the last dose of the investigational drug;
9. Have the ability to give informed consent, have signed informed and able to comply with the treatment plan to visit the tests and other procedural requirements；

Exclusion Criteria:

1. Inadequately treated central nervous system metastases or the presence of uncontrolled or symptomatic active central nervous system metastases；
2. Subjects with peripheral neuropathy；
3. Have received anti-cancer treatment within 4 weeks prior the first dose of study treatment;
4. Are participating in another clinical study or have received the last dose in a clinical study less than 4 weeks from the first dose;
5. Subjects who have received systemic immunosuppressant treatment within 14 days prior the first dose of study treatment;
6. Have received treatment with strong CYP3A inducers or inhibitors, or P-gp inhibitors or inducers within 5 half-lives prior to the first dose;
7. Toxicity and/or complications of previous antitumor therapy has not resolved to NCI-CTCAE level ≤1 or exclusion criteria；
8. Have the following lung diseases or medical history: (1) known or suspected interstitial lung disease; (2) moderate to severe lung diseases that seriously affect lung function within the past 3 months; (3) any autoimmune, connective tissue, or inflammatory disease involving the lungs; (4) prior pneumonectomy; (5) Grade ≥ 3 interstitial lung disease during prior treatment with immune checkpoint inhibitors.
9. Stage 2: ≥ grade 3 immune-related adverse events occurred during previous treatment with immune checkpoint inhibitors；
10. Have any active, known or suspected autoimmune diseases;
11. Moderate or severe ascites with clinical symptoms, uncontrolled or moderate or above pleural effusion and pericardial effusion；
12. The presence of clinical cardiac symptoms or diseases that are not well controlled；
13. Known hereditary or acquired hemorrhage and thrombophilia；
14. Have untreated active hepatitis；
15. Subjects who had a severe infection within 30 days prior to the first dose；
16. Any other malignancy diagnosed within the previous 5 years；
17. Patients with active tuberculosis infection within 1 year prior to enrollment, or with a history of active tuberculosis infection more than 1 year prior but without formal treatment；
18. History of immune deficiency；
19. Live attenuated vaccines were used within 28 days prior to initial study administration or during the expected study period；
20. Known severe allergic reactions to any component of SHR-4602, or other monoclonal antibody/fusion protein drugs；
21. Female subjects who are pregnant or plan to become pregnant during the study period；
22. The presence of uncontrolled mental illness and other conditions known to affect the completion of the study process, such as alcohol, drug or substance abuse, and criminal detention；
23. In the investigator's judgment, there are any other circumstances that may increase the risk of participating in the study, interfere with the study results, or make participation in the study inappropriate.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-12 (Estimated); Primary Completion 2027-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
ORR by investigator assessment | Up to approximately 5 years;
  ORR by investigator assessment was defined as the percentage of participants with confirmed complete response (CR) or partial response (PR), Up to approximately 5 years;

SECONDARY OUTCOMES:
DCR by investigator assessment, | Up to approximately 5 years;
  DCR by investigator assessment was defined as the percentage of participants with confirmed response (CR or PR), or SD, per RECIST v1.1 per investigator, Up to approximately 5 years;
DoR by investigator assessment, | Up to approximately 5 year
  DoR was defined as the time from the first objective response (CR or PR that is subsequently confirmed) to the first documented PD per RECIST v1.1 per investigator or death from any cause, whichever occurs first, Up to approximately 5 years;
PFS by investigator assessment, | Up to approximately 5 years;
  PFS was defined as the time from date of start of study treatment to first documentation of disease progression (PD), or to death due to any cause, whichever occurred first, Up to approximately 5 years;
OS | Up to approximately 5 years;
  OS is defined as the time from start of study treatment to death from any cause, Up to approximately 5 years;
Number of participants with adverse events (AEs), | Up to approximately 5 years;
  An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship, Up to approximately 5 years;

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided